CLINICAL TRIAL: NCT03690622
Title: The Effect of Topical Dexmedetomidine (0.0055%) on Intraocular Pressure in Healthy Eyes: a Randomized Controlled Trial
Brief Title: Effect of Topical Dexmedetomidine on Intraocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beirut Eye Specialist Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeirutEyeSH
Record Dates: First submitted 2018-09-12; First posted 2018-10-01 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Glaucoma; Intraocular Pressure
MeSH Terms: conditions — Glaucoma | interventions — Dexmedetomidine; Hanks Balanced Salt Solution

STUDY DESIGN:
Intervention Model Description: randomised control trial
Who Masked: Participant, Investigator
Masking Description: masking for the drop instilled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSS (Sham Comparator): Balanced salt solution
  Interventions: Drug: Balanced salt solution
- Dexmedetomidine (Active Comparator): dexmedetomidine (0.0055%)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Instillation of eyedrops
  Arms: Dexmedetomidine
Drug: Balanced salt solution — instillation of eyedrop
  Arms: BSS

SUMMARY:
Evaluate the short-term safety and efficacy of dexmedetomidine (0.0055%) drops on intraocular pressure (IOP) in healthy eyes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with healthy eyes and no history of glaucoma

Exclusion Criteria:

* history of glaucoma, IOP > 24mmHg at baseline, abnormal optic nerve on fundus examination, keratoconus, corneal graft, corneal edema or a history of refractive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure change | at presentation, 30 minutes, 4 hours and 24 hours after instillation
  Taken by aplanation tonometry

CONTACTS AND LOCATIONS:
Locations (1):
- Beirut Eye Specialist Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Kim NY, Yoo YC, Park H, Choi YD, Kim CY, Bai SJ. The effect of dexmedetomidine on intraocular pressure increase in patients during robot-assisted laparoscopic radical prostatectomy in the steep Trendelenburg position. J Endourol. 2015 Mar;29(3):310-6. doi: 10.1089/end.2014.0381. Epub 2014 Oct 14. PMID 25137430
- [Background] Zhou C, Zhu Y, Liu Z, Ruan L. The Effects of Intravenous Dexmedetomidine Injections on IOP in General Anesthesia Intubation: A Meta-Analysis. Biomed Res Int. 2017;2017:6186832. doi: 10.1155/2017/6186832. Epub 2017 Feb 2. PMID 28261613
- [Background] Vartiainen J, MacDonald E, Urtti A, Rouhiainen H, Virtanen R. Dexmedetomidine-induced ocular hypotension in rabbits with normal or elevated intraocular pressures. Invest Ophthalmol Vis Sci. 1992 May;33(6):2019-23. PMID 1349879
- [Derived] Fakhoury H, Abdelmassih Y, El-Khoury S, Amro M, Zaarour K, Cherfan C, Tomey K, Khoueir Z. Effect of Topical Dexmedetomidine (0.0055%) on Intraocular Pressure in Healthy Eyes: A Randomized Controlled Trial. J Curr Glaucoma Pract. 2021 May-Aug;15(2):58-63. doi: 10.5005/jp-journals-10078-1310. PMID 34720494
- See also: Patent — http://www.google.com.pg/patents/US8445526